CLINICAL TRIAL: NCT06190743
Title: Perception of Cardiovascular Risk: Description of the Phenomenon in Primary Prevention
Brief Title: Perception of Cardiovascular Risk
Acronym: CV-RP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: IRCCS San Raffaele (Other); Centro Cardiologico Monzino (Other); Istituto Auxologico Italiano (Other); Istituti Ospedalieri Bergamaschi Srl (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.Card.23.01
Record Dates: First submitted 2023-11-27; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Adult individuals who voluntarily wish to participate in prevention events organized by participating centers
  Interventions: Other: Prevention events organized by participating centers

INTERVENTIONS:
Other: Prevention events organized by participating centers — Cardiovascular disease primary prevention events organized by centers participating in the study where capillary sampling will be performed on subjects to quantify plasma levels of cardiovascular risk factors and validated questionnaires will be administered

SUMMARY:
The aim of the study is to describe the association between the perception of cardiovascular (CV) risk and the actual CV risk and, secondarily, to detect the actual CV risk to assess the prevalence of clinical risk factors, determined by means of appropriate instruments.

DETAILED DESCRIPTION:
Cardiovascular (CV) disease is the major cause of premature death in adults that carries serious economic consequences.

Risk perception for CV disease has been reported as the subjective judgment of the likelihood of having a CV event. Risk perception is an important precursor to adopting a healthy lifestyle. However, both overestimation and underestimation of actual risk due mostly to poor health literacy are common.

For these reasons, CV prevention services of health care professionals (e.g., nurses, physicians) should, on the one hand, include screening for the presence of risk factors, and on the other hand, know the CV risk perceptions of those being cared for.

The aim of the study is to describe the association between the perception of cardiovascular (CV) risk, investigated by means of the Perception of Risk of Heart Disease Scale and a Likert-5 scale question, and the actual CV risk according to the SCORE2 and, secondarily, to detect the actual CV risk ascertained by the SCORE2 and to assess the prevalence of clinical risk factors (alterations in the lipid, glucose, or anthropometric profile) determined by means of appropriate instruments.

ELIGIBILITY:
Inclusion Criteria:

* an age between 18 and 69 years of age
* subscription to informed consent.

Exclusion Criteria:

* patients with a positive history of hospitalization due to CV pathology at the time of enrollment;
* patients with ongoing relevant cognitive debilitation (Six Item Screener score < 4)

Ages: 18 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Convenience sample of adult subjects who voluntarily wish to participate in prevention events and who will be asked for consent to participate
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Perception of Risk of Heart Disease Scale | Screening
  Individual perception of the likelihood of having heart disease
Systemic Coronary Risk Estimation version2 | Screening
  Individual real risk at 10 years, both for fatal CV events, and also for nonfatal CV events (myocardial infarction and stroke) in apparently healthy subjects
Patient Health Questionnaire-4 | Screening
  Screening for the uptake of psychological symptoms of anxiety or depression in the primary care setting
Duke-UNC Functional Social Support Questionnaire | Screening
  Strength of affective support derived from people close to the enrolled subjects

SECONDARY OUTCOMES:
Lipid panel | Screening
  Lipid panel measurement
Glucose | Screening
  Glucose measurement
Height | Screening
  Height measurement
Weight | Screening
  Weight measurement

CONTACTS AND LOCATIONS:
Overall Officials: Niccolò Simonelli, Study Nurse, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo
Locations (1):
- Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont, Italy

REFERENCES:
- [Derived] Simonelli N, Alberti M, D'andrea M, Trenta AM, Bagnato E, Faini A, Werba JP, Gianfranceschi E, Rosa D; CV-RP Study Group* on behalf of the Italian Society of Cardiology and in collaboration with the Working Group of Nursing and Technical Care in Cardiology. Correctness of Cardiovascular Risk Perception in Primary Prevention Care: A Multicenter Cross-sectional Italian Study. J Cardiovasc Nurs. 2025 Jul 24. doi: 10.1097/JCN.0000000000001240. Online ahead of print. PMID 40702594